CLINICAL TRIAL: NCT03919682
Title: Promoting Early Detection of Breast Cancer in Rural Rwanda: Impact of a Community Health Worker and Health Center Nurse Training Program
Brief Title: Promoting Early Detection of Breast Cancer in Rural Rwanda: Impact of Community Health Worker and Nurse Training
Acronym: BCED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Breast Cancer Research Foundation (Other); University of Pennsylvania (Other); Partners in Health (Other); Ministry of Health, Rwanda (Other Government)
Responsible Party: Principal Investigator, Lydia Pace, MD, MPH, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014P002688
Record Dates: First submitted 2019-04-12; First posted 2019-04-18 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: early detection; Rwanda
MeSH Terms: conditions — Breast Neoplasms | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training, Phase 1 (Experimental): Community health workers and nurses affiliated with 7 health centers received the breast cancer early detection trainings in April-May 2015
  Interventions: Other: Experimental: Training, Phase 1
- Training, Phase 2 (Experimental): Community health workers and nurses affiliated with 7 health centers received the breast cancer early detection trainings in November-December 2015
  Interventions: Other: Experimental: Training, Phase 2
- Control (No Intervention): 6 health centers served as controls and did not receive training during the study period

INTERVENTIONS:
Other: Experimental: Training, Phase 1 — Weeklong training in signs, symptoms and treatability of breast cancer, performance of clinical breast exam, and structured algorithms for management of breast complaints followed by regular mentorship for health center nurses. CHWs received a one-day training in breast awareness and how to educate communities about breast health.
  Arms: Training, Phase 1
Other: Experimental: Training, Phase 2 — Weeklong training in signs, symptoms and treatability of breast cancer, performance of clinical breast exam, and structured algorithms for management of breast complaints followed by regular mentorship for health center nurses. CHWs received a one-day training in breast awareness and how to educate communities about breast health.
  Arms: Training, Phase 2

SUMMARY:
This project proposes a pilot intervention in Burera District to train rural Rwandan community health workers (CHWs) in breast awareness, and to train primary care nurses at rural health centers in the assessment and management of breast complaints, with a focus on when patients must be urgently referred for more advanced evaluation. The project will randomize health centers to receive the intervention and will evaluate the impact of these trainings on nurse and CHW knowledge and skills. In order to help Rwanda prepare for national early detection efforts, the investigators will also assess the impact of these trainings on patient volume at the health center level, and visits and further diagnostic testing at the district hospital level. The investigators will also examine the impact on the length of diagnostic delays experienced by patients with a breast problem. Among those patients diagnosed with breast cancer, the investigators will also assess their stage at diagnosis.

ELIGIBILITY:
Inclusion Criteria

* Community health workers or health center nurses affiliated with a designated intervention health center
* Interested in participating

Exclusion Criteria

* Not interested in participating
* Not available for training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1203 (Actual)
Dates: Start 2015-04-18 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2017-04-17 (Actual)

PRIMARY OUTCOMES:
Health center nurse knowledge | up to 6 months
  Nurses' knowledge will be assessed through written tests administered immediately before and immediately after trainings, and delayed post-tests administered 3 to 6 months after training. The investigators will use an adapted instrument that incorporates the Breast Cancer Knowledge Test and other surveys to assess clinician knowledge about breast cancer risk, signs and symptoms, and treatability. Questions were developed through review of existing instruments used in the United States, Mexico, the United Kingdom, and Nigeria, and expert input, feedback from clinical colleagues in Rwanda, and pilot testing with Rwandan hospital-based nurses. We will assess each nurse's overall test score as the total percentage of questions correct and assess scores within specific knowledge domains. The more questions answered correctly and the higher the score, the better the outcome (the score represents the percent of questions answered correctly).
Community health worker knowledge | up to 6 months
  CHWs' knowledge will be assessed through written tests administered immediately before and immediately after trainings, and delayed post-tests administered 3 to 6 months after training. The investigators will use an adapted instrument that incorporates the Breast Cancer Knowledge Test and other surveys to assess clinician knowledge about breast cancer risk, signs and symptoms, and treatability. Questions were developed through review of existing instruments used in the United States, Mexico, the United Kingdom, and Nigeria, and expert input, feedback from clinical colleagues in Rwanda, and pilot testing with Rwandan hospital-based nurses. We will assess each CHW's overall test score as the total percentage of questions correct and assess scores within specific knowledge domains. The more questions answered correctly and the higher the score, the better the outcome (the score represents the percent of questions answered correctly).
Health center nurse clinical skills | up to 16 months
  Nurses' performance scores on clinical breast exam checklists that assess completion of the steps required for high-quality clinical breast exam and are based on other published checklists adapted to the rural Rwandan setting. CBE materials were based on CBE guidelines and published and unpublished curricula adapted to our setting. During her regular health center visits, the breast health mentor will assess nurses' clinical skills in their clinics by using a checklist that includes the same questions as the pre- and post-test assessment form. When possible, the mentor will assess individual nurses by using the same checklist two or more times during a given clinical session, including one at the beginning of a session. We will analyze checklists completed between May 2015 and September 2016. The more actions performed correctly and the higher the score, the better the outcome (the score represents the percent of actions performed correctly).

SECONDARY OUTCOMES:
Health center volume | 30 months
  Number of patients per month with breast concerns presenting at health centers before versus after the intervention, and compared with control health centers.
District hospital referrals | 30 months
  Number of patients from intervention health centers requiring referral to the district hospital before versus after the intervention, and compared with patients from control health centers.
Breast ultrasounds | 30 months
  Number of patients from intervention health centers requiring ultrasound before versus after the intervention, and compared with patients from control health centers
Breast biopsy | 30 months
  Number of patients from intervention health centers requiring breast biopsy before versus after the intervention, and compared with patients from control health centers.
Patient delays | 24 months
  Among patients referred from intervention versus control health centers to the hospital for breast concerns, length of time experienced between onset of symptoms and first presentation to a health center.
System delays | 24 months
  Among patients referred from intervention versus control health centers to the hospital for breast concerns, length of time experienced between first presentation at a health center and first presentation at the hospital.
Breast cancer detection rate | 30 months
  Among patients referred to the hospital from intervention health centers, proportion diagnosed with breast cancer compared to the proportion among those referred from control health centers, and the proportion from intervention health centers before the trainings.
Breast cancer stage | 30 months
  Among patients diagnosed with breast cancer from intervention health centers, the AJCC versus 7 clinical breast cancer stage documented in hospital medical records. The investigators will compare the proportion of patients presenting with Stage I or II stage disease to the proportion with stage I or II disease among those referred from control health centers, and those from intervention health centers before the trainings.